CLINICAL TRIAL: NCT03202914
Title: Metabolomics for Identifying Biomarkers of Dietary Intake and Kidney Disease Progression: A Secondary Data Analysis of the Modification of Diet in Renal Disease (MDRD) Study
Brief Title: Metabolomics for Identifying Biomarkers of Dietary Intake and Kidney Disease Progression
Acronym: MDRD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Tufts Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB00007383; K01DK107782 (NIH)
Record Dates: First submitted 2017-06-23; First posted 2017-06-29 (Actual); Last update posted 2017-06-29 (Actual); Status verified 2017-06

CONDITIONS: Dietary Modification; Kidney Diseases, Chronic
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Diet, Protein-Restricted; Phosphorus

STUDY DESIGN:
Intervention Model Description: The present study consists of a secondary data analysis of the MDRD Study. Planned analyses will be limited to participants with available stored specimens.
  The original MDRD Study was a 2 x 2 factorial study design, in which individuals were randomized to amounts of protein and phosphorus intake and levels of blood pressure control. In this secondary data analysis, we will analyze metabolites according to level of protein intake and will adjust for the blood pressure intervention.
Who Masked: Outcomes Assessor
Masking Description: During the original MDRD Study, clinical center personnel as well as study participants were masked to the results of the outcome assessment during the follow-up period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Usual protein and phosphorus diet (Active Comparator): protein: 1.3 g/kg/day, phosphorus: 16-20 mg/kg/day
  Interventions: Behavioral: Usual protein and phosphorus diet
- Low protein and phosphorus diet (Active Comparator): protein: 0.58 g/kg/day with ≥0.35 g of protein high in amino acids, phosphorus: 5-10 mg/kg/day
  Interventions: Behavioral: Low protein and phosphorus diet
- Very low protein and phosphorus (Experimental): protein: 0.28 g/kg/day, phosphorus: 4-9 mg/kg/day; keto-acid and amino acid supplement (0.28 g/kg/day)
  Interventions: Behavioral: Very low protein and phosphorus

INTERVENTIONS:
Behavioral: Usual protein and phosphorus diet — Diet intervention
  Arms: Usual protein and phosphorus diet
Behavioral: Low protein and phosphorus diet — Diet intervention
  Arms: Low protein and phosphorus diet
Behavioral: Very low protein and phosphorus — Diet intervention
  Arms: Very low protein and phosphorus

SUMMARY:
The present record represents a secondary data analysis of the Modification of Diet in Renal Disease (MDRD) Study. For this analysis, the MDRD study data and specimens were retrieved from the National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) Central Repository. A global, untargeted, metabolomic profile was used to investigate biomarkers of dietary intake as well as biomarkers of kidney disease progression.

DETAILED DESCRIPTION:
The present study was conducted in order to: 1) quantify the metabolomic expression of dietary intake; and 2) examine the relationship between metabolites that reflect dietary intake and kidney disease progression. This secondary data analysis leverages the completed Modification of Diet in Renal Disease (MDRD) study, a randomized clinical trial of dietary protein restriction (N=840).

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70
* Evidence of chronic renal disease with increased serum creatinine (men: 1.4-7.0 mg/dL, women: 1.2-7.0 mg/dL)
* Mean arterial blood pressure less than or equal to 125 mmHg

Exclusion Criteria:

* Insulin-dependent diabetes
* Kidney transplant recipient

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 840 (Actual)
Dates: Start 1988-10 (Actual); Primary Completion 1993-05 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Serum metabolomic profile | 12 month follow-up visit
  Metabolites were measured using a global, untargeted, metabolomic platform in serum specimens collected at the 12 month follow-up visit in the MDRD Study. Reverse phase, untargeted ultra-performance liquid chromatography tandem mass spectrometry quantification was used to measure metabolites. Peaks were quantified by calculating the area under the curve. Data were normalized to account for day-to-day instrumental variation. Compounds were identified by comparison to a library of purified standards or recurrent unknown entities and matches were determined based on retention time, mass-to-charge ratio, and chromatographic data.

CONTACTS AND LOCATIONS:
Overall Officials: Casey M. Rebholz, PhD, MPH, MS, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Johns Hopkins Bloomberg School of Public Health, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Levey AS, Adler S, Caggiula AW, England BK, Greene T, Hunsicker LG, Kusek JW, Rogers NL, Teschan PE. Effects of dietary protein restriction on the progression of advanced renal disease in the Modification of Diet in Renal Disease Study. Am J Kidney Dis. 1996 May;27(5):652-63. doi: 10.1016/s0272-6386(96)90099-2. PMID 8629624
- [Result] Klahr S, Levey AS, Beck GJ, Caggiula AW, Hunsicker L, Kusek JW, Striker G. The effects of dietary protein restriction and blood-pressure control on the progression of chronic renal disease. Modification of Diet in Renal Disease Study Group. N Engl J Med. 1994 Mar 31;330(13):877-84. doi: 10.1056/NEJM199403313301301. PMID 8114857
- [Derived] Rebholz CM, Zheng Z, Grams ME, Appel LJ, Sarnak MJ, Inker LA, Levey AS, Coresh J. Serum metabolites associated with dietary protein intake: results from the Modification of Diet in Renal Disease (MDRD) randomized clinical trial. Am J Clin Nutr. 2019 Mar 1;109(3):517-525. doi: 10.1093/ajcn/nqy202. PMID 30753252